CLINICAL TRIAL: NCT06886386
Title: Effects of Trans-spinal Direct Current Stimulation Combined to Physical Therapy in Patients with Chronic Incomplete Spinal Cord Injury
Brief Title: TsDCS and Physical Therapy After Incomplete Spinal Cord Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Fernanda Natacha Rufino Nogueira, Master in Physical Therapy, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tsDCS_physical therapy_iSCI
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury
Keywords: trans-spinal direct current stimulation; physical therapy; spinal cord injury; motor function
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tsDCS + physical therapy (Experimental): a randomized, sham-controlled, double-blinded and parallel group trial (10 therapeutic sessions) with the combination between physical therapy combinated and active tsDCS in improving the motor function of adult patients with chronic incomplete spinal cord injury. The sessions will be performed five times a week for a month.
  Interventions: Device: Trans-spinal direct current stimulation
- sham tsDCS + physical therapy (Sham Comparator): a randomized, sham-controlled, double-blinded and parallel group trial (10 therapeutic sessions) with the combination between physical therapy combinated and sham tsDCS in improving the motor function of adult patients with chronic incomplete spinal cord injury. The sessions will be performed five times a week for a month.
  Interventions: Device: Trans-spinal direct current stimulation

INTERVENTIONS:
Device: Trans-spinal direct current stimulation — Patients with a neurological level above T10 will receive cervical tsDCS (anode electrode at C7, and the cathode electrode on the right shoulder). Patients with a neurological level from T10 onwards will receive thoracic tsDCS (anode electrode at T10, and the cathode electrode at the iliac crest). (i) Experimental group (active tsDCS): electrical stimulator (Neuroconn/Germany) connected to a pair of saline-soaked sponge electrodes (35 cm²) with a current intensity of 2.5 mA for 20 minutes. (ii) Control group (sham tsDCS) with electrodes positioned at the same locations as active tsDCS, for 30 seconds (the setup will remain for the full 20 minutes). Thus, patients will experience the initial sensations at the stimulated site, without inducing an effect. Physical therapy will be performed during tsDCS (45 minutes), based on scientific evidence, considering patient preferences, and respecting motor learning theory and neuroplasticity principles, focusing on motor function recovery.
  Other Names: Physical therapy

SUMMARY:
The aim of this study is to evaluate the effects of tsDCS combined with physical therapy on the recovery of motor function in adult patients with chronic incomplete spinal cord injury.

DETAILED DESCRIPTION:
A randomized, sham-controlled, double-blinded and parallel group trial (10 therapeutic sessions). Active or sham tsDCS will be combined with physical therapy to verify the improvement of motor function in patients with incomplete spinal cord injury. Assessments will be performed before and after therapeutic sessions and at the 30-day follow-up after the intervention, through: (i) ASIA Lower and Upper Extremities Motor Scale (LEMS and UEMS), (ii) ASIA Impairment Scale (AIS), (iii) Ashworth Modified Scale; (iv) the Functional Independence Measure (SCIM-III), and (v) the Patient Global Impression of Change Scale - (PGICS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of incomplete spinal cord injury by a neurologist
* Diagnosis time greater than 12 months

Exclusion Criteria:

* Patients with additional current neurological diagnoses
* Presence of contraindications for tsDCS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Changes in the Upper and Lower Extremities Motor Scale (UEMS and LEMS) from ASIA. | Before the sessions, after 10 sessions (10 days of intervention) and one month (30 days) following the completion of the study.
  It is an international scale. The UEMS and LEMS are composed of the sum of muscle function grading for the five key muscles of the upper and lower limbs (respectively) as defined by ASIA. The score for each muscle is graded from '0' to '5', and the total score can range from '0' to '50'. To calculate this, the scores for the five muscles of each limb (upper and lower/ left and right) should be summed. The higher the score, the better the motor function.

SECONDARY OUTCOMES:
Changes on American Spinal Cord Injury Association - Impairment Scale (AIS) | Before the sessions, after 10 sessions (10 days of intervention) and one month (30 days) following the completion of the study.
  This is international scale, it is the gold standard for the diagnosis of spinal cord injury and is used worldwide. The AIS categorizes the lesion from full spinal cord injury to normal degree (severity of the injury), according to sensory-motor preservation, passing through degrees of spinal cord injury (A , B, C, D or E).
  (i) AIS A (Complete): no motor or sensory function preserved in the sacral regions (S4-S5); (ii) AIS B (Sensory incomplete): sensory function, but not motor, preserved below the neurological level; (iii) AIS C (Motor incomplete): motor function preserved, with more than half of the muscles scoring less than 3; (vi) AIS D (Motor incomplete): motor function preserved, with more than half of the muscles scoring 3 or more; and (v) AIS E (Normal): normal motor and sensory function. Observations: "AIS A" represents the worse outcome regarding the severity of the injury, and "AIS E" represents the better.
Changes on Spinal cord independence measure (Self-Reported) III (SCIM-III) | Before the sessions, after 10 sessions (10 days of intervention) and one month (30 days) following the completion of the study.
  The scale assesses patients' ability to perform tasks inherent to spinal cord injury and detects improvements in their functionality. The SCIM-III is a scale from 0 to 100 points and divides into three main domains: self-care (feeding, bathing, dressing and cleanliness), breathing, sphincter control and mobility (indoors and out home and transfers). Higher scores on the SCIM III reflect higher levels of independence.
Change from Modified Ashworth scale (MAS) | Before the sessions, after 10 sessions (10 days of intervention) and one month (30 days) following the completion of the study.
  The Modified Ashworth Scale is a clinical measure for assessing muscle tone during passive movement with speed dependence and shows good validity and reproducibility. In this study, it will assess the following muscles: hip flexors and extensors, knee flexors and extensors, ankle dorsiflexors and plantar flexors; shoulder flexors and extensors, elbow flexors and extensors, wrist flexors and extensors. The instrument categorizes spasticity into six different grades, ranging from "0" (normal muscle tone) to "4" (joint rigidity in flexion or extension). The lower the score, the less spasticity assessed.
Changes on Patient Global Impression of Change Scale - (PGICS) | After 10 sessions (10 days of intervention) and one month (30 days) following the completion of the study.
  The PGICS is a one-dimensional measure in which individuals rate their improvement associated with intervention on a scale of 7 items ranging from "1 = no change" to "7 = Much better". This scale has already been validated in Brazil and has been used in clinical practice assays with spinal cord injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil